CLINICAL TRIAL: NCT02401061
Title: A Phase 1/2, Open-Label, Dose Escalation Study of PRTX-100 in Adult Patients With Persistent/Chronic Immune Thrombocytopenia
Brief Title: PRTX-100-202 Open-Label, Dose Escalation Study in Adult Patients With ITP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enough data has been collected to allow analysis of safety profile and risk-benefit.
Sponsor: Protalex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRTX-100-202
Record Dates: First submitted 2015-03-18; First posted 2015-03-27 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — Staphylococcal Protein A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRTX-100 (Experimental): Patients will be assigned to consecutive PRTX-100 interventions as they are enrolled into the study. Between two and six patients will be enrolled per intervention level. Intervention levels range from one (1) to twenty four (24) micrograms of PRTX-100 per kilogram of patient weight. Patients may receive up to four weekly infusions of PRTX-100 over the study treatment period. PRTX-100 doses ≤ 500 μg will be infused intravenously over 30 minutes. PRTX-100 doses > 500 μg will be infused over 60 minutes. Patients will remain under observation for 4 hours after completion of PRTX-100 dosing for safety management.
  Interventions: Drug: PRTX-100

INTERVENTIONS:
Drug: PRTX-100 — Four weekly infusions of PRTX-100 at a level of 1 (3, 6,12, 18, or 24) microgram of PRTX-100 per kilogram of patient weight, infused over 30 minutes, followed by four hours of observation.
  Other Names: SpA; Staphylococcal Protein A

SUMMARY:
Pre-clinical and clinical evaluations show that PRTX- 100 has biological activity that may lead to improved platelet levels where these are decreased due to immunological pathologies and that PRTX-100 has an acceptable safety profile. In vivo treatment with PRTX-100 has been shown to raise platelet counts in a mouse model of immune thrombocytopenia (ITP). The primary objective of the study is to assess the efficacy of PRTX-100 in terms of platelet response in patients with chronic/persistent ITP.

Funding Source - FDA OOPD (1R01FD005750-01A1)

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to initiation of any study-related procedures
2. Male or female ≥ 18 years of age
3. ITP that has persisted for ≥ 3 months. ITP must be diagnosed in accordance The American Society of Hematology 2011 Evidence-based Practice Guideline for Immune Thrombocytopenia (Neunert et al. 2011) or the International Consensus Report on The Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as locally applicable.
4. Received ≥ 1 typical regime for the treatment of ITP. Splenectomy is considered one standard ITP treatment
5. A mean platelet count of < 30,000/μL, with no individual platelet count > 35,000/μL; or for those subjects receiving a constant dose of permitted treatments for ITP: a mean platelet count < 50,000/μL, with no count greater than 55,000/μL. (Note: The mean platelet count must be determined based on 2 platelet counts including one obtained within ≤ 7 days of first PRTX-100 dose and the other within ≤ 30 days of the first dose of PRTX-100.)
6. If on corticosteroids, a dose of < 1 mg/kg prednisone per day or equivalent that has been stable for ≥ 21 days prior to the first dose of PRTX-100. High-dose pulse steroid therapy is NOT allowed within 14 days prior to the first dose of PRTX-100.
7. If receiving eltrombopag or romiplostim, the dose must have been stable for ≥ 21 days prior to the first dose of PRTX-100
8. If on steroid-sparing adjunctive immunosuppression with cyclosporine, azathioprine, mycophenolate, or 6-mercaptopurine, the dose must have been stable for ≥ 30 days prior to the first dose of PRTX-100 and must be expected to remain stable through study Day 29, unless dose reduction is required due to toxicities. Treatment with other cytotoxic agents (e.g. cyclophosphamide, vincristine) are not allowed within three months prior to the first dose of PRTX- 100.
9. Any prior treatment with rituximab or any other anti-CD20 agent must have been > 6 months prior to the first dose of PRTX-100
10. If female, must not be pregnant (pregnancy testing will be performed locally in all female patients of childbearing potential), must not be nursing and must be one of the following:

    * Surgically sterile (bilateral tubal ligation, hysterectomy)
    * Postmenopausal with last natural menses > 24 months prior
    * Premenopausal and using an acceptable form of birth control. Acceptable forms of birth control include: hormonal contraceptives (implantable, oral, patch) used for ≥ 2 months prior to screening or double barrier methods (any combination of two of the following: intrauterine device [IUD], male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). All premenopausal females must have a negative urine or serum pregnancy test at screening and on Day 1 prior to first PRTX-100 treatment.

Exclusion Criteria:

1. Splenectomy ≤ 90 days prior to the first dose of PRTX-100
2. Unstable coronary artery disease or other medical condition (such as type 1 diabetes) that, in the Investigator's opinion, might increase the risk to the patient
3. Evidence of active infection requiring antibiotic therapy ≤ 14 days prior to the first dose of PRTX- 100
4. Myelodysplastic syndrome. If clinically significant anemia or pancytopenia exists, documentation of a bone marrow aspirate within 24 months prior to the first dose of PRTX-100 showing no evidence of myelodysplasia is required.
5. Medical history of vasculitis or lupus erythematosus
6. Propensity to allergic reactions defined as a history of allergic reaction to more than one medication
7. History of any treatment for cancer within the past two years other than basal cell or squamous cell carcinoma of the skin that has been treated with curative intent
8. Seropositive for human immunodeficiency virus (HIV)
9. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B or C (positive for hepatitis B surface antigen or positive anti-hepatitis C antibody test) and evidence of current or active infection (e.g. HCV RNA test)
10. History suggestive of substance abuse
11. History or evidence on physical examination or screening laboratory tests of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the study drug
12. Treatment with IVIG ≤ 14 days prior to the first dose of PRTX-100
13. Treatment with an anti-Rh D antigen agent (e.g. WinPho) ≤ 14 days prior to the first dose of PRTX-100
14. Use of any investigational drug, other than eltrombopag or romiplostim, ≤ 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the first dose of RTX-100
15. Not willing to stay at the study site for 4 hours after each PRTX-100 infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2019-03 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Platelet Response, Change from Baseline | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The primary efficacy endpoint is platelet response defined as a platelet count ≥ 30,000/μL and at least a doubling of baseline platelet count (determined on Day 1 prior to PRTX-100 administration) in patients with a baseline platelet count < 30,000/μL. In patients receiving permitted treatments for ITP with a baseline platelet count ≥ 30,000/μL and < 50,000/μL, an increase in platelet count to ≥ 50,000/μL and at least a doubling of baseline platelet count or an increase to > 100,000/μL be considered a platelet response.

SECONDARY OUTCOMES:
Complete platelet response, Change from Baseline | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  Defined as a platelet count ≥ 100,000/μL
Time to platelet response defined as the mean number of days from first PRTX-100 dose until platelet response | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The mean number of days from first PRTX-100 dose until platelet response
Durability of platelet response | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  The number of days from first documented platelet response to first platelet count below platelet response criteria
Concomitant ITP medication use (frequency and amount) | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  ITP medications include eltrombopag, romiplostim, steroid-sparing adjunctive treatment (e.g. cyclosporine, azathioprine, mycophenolate, danazol, dapsone, or 6-mercaptopurine), and any ITP rescue medications (e.g. IVIG) received during the study Screening and Treatment Periods
Adverse Events | Days 3, 8, 15, 22, 29, 36, 43, 50, 78, 106, 169, and 337
  Safety will be described by AEs, SAEs, infusion reactions, clinical laboratory tests (hematology, blood chemistry and urinalysis), vital signs, physical findings and ECGs. AE severity will be graded according to Toxicity Grading Criteria derived from published standards

CONTACTS AND LOCATIONS:
Overall Officials: William E Gannon Jr., MD, Study Director — Protalex, Inc.
Locations (11):
- United States (6):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Weil-Cornell Medical College, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen, AB
  - Leicester Royal Infirmary, Leicester, Leichester
  - Queen Elizabeth Hospital, Birmingham
  - Glasgow Royal Infirmary, Glasgow
  - Norfolk and Norwich Hospital, Norwich